CLINICAL TRIAL: NCT04239846
Title: A Randomized, Double-blind, Placebo-controlled Trial of AC-701 for Treatment of Skin Rash in Subjects With EGFR Inhibitor Therapy
Brief Title: Prophylactic Treatment of Skin Rash Associated With EGFR Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AC-701-ONC-002
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: EGFR Inhibitor-Induced Skin Rash

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AC-701 (Experimental): AC-701 Topical Gel 0.3%
  Interventions: Drug: AC-701 Topical Gel 0.3%
- Placebo (Placebo Comparator): Placebo Gel
  Interventions: Other: Placebo Gel

INTERVENTIONS:
Drug: AC-701 Topical Gel 0.3% — AC-701 Topical Gel 0.3%, BID
  Other Names: AC-701
  Arms: AC-701
Other: Placebo Gel — Placebo Gel, BID
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
Epidermal growth factor receptor inhibitor (EGFRI) therapy for cancer is associated with potentially severe face and trunk skin acneiform rash. Severe or persistent side effects may lead to decreased dose, interruption or discontinuation of EGFRI treatment. Inflammation is believed to play an important role in EGFRI-induced skin toxicity as a number of proinflammatory cytokines induced by EGFRI are released from epidermal cells, resulting in activation and recruitment of immune cells such as neutrophils and lymphocytes, and subsequent development of skin reaction associated with keratinocyte apoptosis. AC-701 has been reported its antibiotic and anti-inflammatory activities in literature, and further demonstrated in vitro effect to prevent the secretion of inflammatory cytokines associated with EGFR inhibition. This study is to evaluate the prophylactic efficacy of topical AC-701 in subjects with skin rash associated with EGFRI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Is between 20 and 80 years of age, inclusive.
2. Patients who are within ±3 days of initiating EGFR inhibitor therapy using afatinib or erlotinib, and have no prior history of using afatinib or erlotinib within 6 months.
3. Has a life expectancy of at least three months.

Exclusion Criteria:

1. Has any active dermatological conditions of the face that may interfere with the diagnosis, assessment, or treatment of face skin rash associated with targeted cancer therapy.
2. Has been treated with steroids (systemic or topical on face) to the face within 7 days prior to Day 1.
3. Patients who have been treated with oral antibiotics that known to exert anti-inflammatory effect (such as doxycycline or minocycline) within 7 days prior to Day 1.
4. Is currently treated with target therapy other than afatinib or erlotinib.
5. Receive prior treatment with any investigational product within 28 days prior to Day 1.
6. Has hypersensitivity or allergy to the study medication.
7. Has any other significant diseases, conditions, or laboratory values which, in the opinion of the investigator, might make participation not in the subject's best interest or confound the interpretation of study results.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Number of subjects with MESTT Grade 0 or 1 | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Emily Lin, Study Director — TWi Biotechnology, Inc.
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No